CLINICAL TRIAL: NCT06442683
Title: Efficacy of Simulation-based Neonatal Echocardiography Training: a Randomized Controlled Trial
Brief Title: Efficacy of Simulation-based Neonatal Echocardiography Training (SimuEchoNeo)
Acronym: SimuEchoNeo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ID2259
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Simulation-based Training on Residents
Keywords: Neonatology; Simulation-based training; Echocardiography

STUDY DESIGN:
Intervention Model Description: Multicentered randomized controlled trial.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation group (Experimental): Theorical training, simulation-based training and bedside training
  Interventions: Diagnostic Test: TTE simulation-based medical training
- Control group (No Intervention): Theorical and bedside training

INTERVENTIONS:
Diagnostic Test: TTE simulation-based medical training — half-day simulation-based neonatal echocardiography training.
  Arms: Simulation group

SUMMARY:
Echocardiographic examination plays a critical role in neonatology, but its bedside training faces challenges due to limited patient access. While simulation training has proven effective in different fields of adult medical care, its application in neonatal echocardiography remains unexplored.

Researchers will compare simulation-based training to usual training (theorical and bedside) for neonatal echocardiography among pediatric residents to see if simulation-trained residents have better skills.

Participants will undergo :

* theorial, simulation-based and bedside training or
* theorical and bedside training only.

DETAILED DESCRIPTION:
All participants were granted full access to the online theorical course throughout the semester of participation, which encompass a presentation of the study and a theorical training. In addition, during their Neonatal Intensive Care Unit (NICU) residency/night shifts, all residents had the possibility to learn bedside transthoracic echocardiography (TTE) and document their experiences using a collection form provided at the time of inclusion.

Beyond access to the e-learning, the simulation group participated in standardized training using the neonatal simulator EchoCom|Neo during the first month of their 6-month residency in NICU. The training session involved a maximum of four residents at the same time, one teacher and one EchoCom|Neo simulator.

The session consisted of the modified Peyton 4-steps process (demonstration, deconstruction, comprehension, performance) with the normal heart scenario set on the simulator, presentation of a persistent ductus arteriosus (PDA), a pericardial effusion case and an evaluation of each resident individually, on the simulator set with normal heart scenario, performing a TTE with a description of the visible structures. The minimum passing score for the validation of the training session was set at 12 out of 14 (reference score, table 1). If the minimum passing score was not achieved, a second training session must have been scheduled until the minimum passing score was reached.

The entire simulation session typically lasted between 2.5 to 3 hours. For standardization of training sessions, pre-registered videos were used whenever applicable (presentation of the simulation session, presentation of the simulator, and first and second Peyton's steps), and the training was conducted by the same teacher throughout the study, in the respective hospital of each resident (Caen, Rouen or Tours).

Two evaluation timepoints were defined at the middle (3 to 4 months after initial training, M3-M4), and at the end of the 6-month residency (6 months after the training, M6).

The evaluation session took place using the EchoCom|Neo simulator (EchoCom GmbH, Nieheim, Germany), set with the normal heart scenario, and placed on an open neonatal warmer, in the respective hospital of each resident. Each resident was evaluated individually with video recording for second evaluation.

Before starting the evaluation, each resident had 5 minutes to familiarize themselves with the handling of the simulator probe. They were asked to perform 7 TTE sections, with the teacher listing each expected TTE section at the beginning of the evaluation.

At each evaluation session, two evaluators conducted independent assessments. One evaluator was a pediatric cardiologist, blinded to the randomization, while the other was a pediatric resident (the simulation TTE training's teacher). One evaluator was physically present during the evaluation, while the other used video recording. Each evaluator assigned two scores for each resident:

* A reference score: 2 points for each section (optimal, suboptimal, not found), total out of 14 points.
* A custom-made score: 1 point for each anatomic structure within each section, emphasizing visualization and recognition of heart structures, total out of 33 points.

The duration of the TTE at 3 and 6 months were also recorded with second precision. Following the second evaluation at M6, the number of bedside TTE performed was documented, and a satisfaction questionnaire based on a Likert scale was requested.

ELIGIBILITY:
Inclusion Criteria:

* residents at all training levels (from first to fifth year) completing a 6-month residency or at least night shifts in neonatology at one of the 3 French NICUs involved (University Hospitals of Caen, Rouen or Tours)

Exclusion Criteria:

* Residents who had already received a TTE training (cardiology or cardiopediatrics 6-month residency or postgraduate training in cardiology or echocardiography)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Transthoracic echocardiography (TTE) score at 3 months | 3 to 4 months after initial training
  Difference in TTE score at 3 months between the two groups

SECONDARY OUTCOMES:
TTE score at 6 months | 6 months after initial training
  Difference in TTE score at 6 months between the two groups
TTE duration | 3-4 months and 6 months
  TTE duration at 3 and 6 months
Satisfaction score at 6 months | 6 months
  Satisfaction score over 25 points

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University Hospital of Caen, Caen
  - University Hospital of Rouen, Rouen
  - University Hospital of Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (including data dictionaries) will be made available, in addition to study protocols, the statistical analysis plan, and the informed consent form. The data will be made available upon publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be submitted to amelie.blanchetiere[at]unicaen.fr.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: when asked.

REFERENCES:
- [Derived] Blanchetiere A, Guillouet E, Favrais G, Lardennois C, Bellot A, Savey B. Simulation-Based Echocardiography Training Enhanced Competence and Self-Confidence in Neonatal Residents. Acta Paediatr. 2025 Jul;114(7):1623-1632. doi: 10.1111/apa.70003. Epub 2025 Jan 31. PMID 39891031